CLINICAL TRIAL: NCT02094612
Title: Effectiveness of the Quotient® ADHD Assessment in a System of Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Pearson/Clinical Assessment (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CN-13-1692-H; Quotient ADHD (Other: Abbreviated study title)
Record Dates: First submitted 2014-03-13; First posted 2014-03-24 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-06

CONDITIONS: Attention Deficit and Disruptive Behavior Disorders; Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit and Disruptive Behavior Disorders; Attention Deficit Disorder with Hyperactivity; Pediatrics; Patient Outcome Assessment
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Active Comparator): Usual clinic ADHD care
  Interventions: Behavioral: Usual Clinic ADHD Care
- Usual Care plus Assessment (Experimental): Usual clinic ADHD care plus the Quotient®
  Interventions: Device: Quotient®

INTERVENTIONS:
Device: Quotient® — Patients will be randomized once at the time of ADHD assessment to either usual clinic ADHD care or usual clinic ADHD care plus the Quotient using computer-generated random numbers.
  Other Names: OpTAX
  Arms: Usual Care plus Assessment
Behavioral: Usual Clinic ADHD Care — Usual ADHD care as provided by the clinic
  Arms: Usual Care

SUMMARY:
The study goal is to examine whether the use of an objective computerized neuroassessment (the Quotient System) for Attention-Deficit/Hyperactivity Disorder (ADHD) is related to improved outcomes among pediatric patients being assessed and treated for ADHD.

DETAILED DESCRIPTION:
This study is a randomized, controlled trial using a 2-phase data collection. The first phase is the initial assessment for ADHD and includes all patients eligible to be assessed for ADHD as determined by their clinician in the course of usual care. The baseline measurements will be used to compare groups at baseline, and also for longitudinal analyses of medication management. Patients are randomized at this point. Patients in both treatment arms who then receive an ADHD diagnosis and who start medication for ADHD will be eligible for the second phase of the study: three follow-up assessments over six months. Patients who do not have an ADHD diagnosis will not continue in the study, and will be treated by their clinician as usual.

ELIGIBILITY:
Inclusion Criteria:

* All patients within the specified age range who are English speaking and who are presenting for ADHD assessment are eligible. An additional criterion is consent to be randomized.

Exclusion Criteria:

* Non English speaking
* Refusal to participate

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 207 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia I Campbell, PhD, Principal Investigator — Kaiser Permanente
Locations (3):
- United States (3):
  - Kaiser Permanente, Folsom, Folsom, California
  - Kaiser Permanente, Roseville, Roseville, California
  - Kaiser Permanente, Walnut Creek Medical Center, Walnut Creek, California

REFERENCES:
- [Background] Chinchilli VM, Fisher L, Craig TJ. Statistical issues in clinical trials that involve the double-blind, placebo-controlled food challenge. J Allergy Clin Immunol. 2005 Mar;115(3):592-7. doi: 10.1016/j.jaci.2005.01.008. PMID 15753909
- [Background] Clinical practice guideline: diagnosis and evaluation of the child with attention-deficit/hyperactivity disorder. American Academy of Pediatrics. Pediatrics. 2000 May;105(5):1158-70. doi: 10.1542/peds.105.5.1158. PMID 10836893
- [Background] Foy JM, Earls MF. A process for developing community consensus regarding the diagnosis and management of attention-deficit/hyperactivity disorder. Pediatrics. 2005 Jan;115(1):e97-104. doi: 10.1542/peds.2004-0953. PMID 15629972
- [Background] Herrerias CT, Perrin JM, Stein MT. The child with ADHD: using the AAP Clinical Practice Guideline. American Academy of Pediatrics. Am Fam Physician. 2001 May 1;63(9):1803-10. PMID 11352293
- [Background] Jensen PS, Garcia JA, Glied S, Crowe M, Foster M, Schlander M, Hinshaw S, Vitiello B, Arnold LE, Elliott G, Hechtman L, Newcorn JH, Pelham WE, Swanson J, Wells K. Cost-effectiveness of ADHD treatments: findings from the multimodal treatment study of children with ADHD. Am J Psychiatry. 2005 Sep;162(9):1628-36. doi: 10.1176/appi.ajp.162.9.1628. PMID 16135621
- [Background] Lachin JM, Foulkes MA. Evaluation of sample size and power for analyses of survival with allowance for nonuniform patient entry, losses to follow-up, noncompliance, and stratification. Biometrics. 1986 Sep;42(3):507-19. PMID 3567285
- [Background] Langberg JM, Froehlich TE, Loren RE, Martin JE, Epstein JN. Assessing children with ADHD in primary care settings. Expert Rev Neurother. 2008 Apr;8(4):627-41. doi: 10.1586/14737175.8.4.627. PMID 18416664
- [Background] Leslie LK, Weckerly J, Plemmons D, Landsverk J, Eastman S. Implementing the American Academy of Pediatrics attention-deficit/hyperactivity disorder diagnostic guidelines in primary care settings. Pediatrics. 2004 Jul;114(1):129-40. doi: 10.1542/peds.114.1.129. PMID 15231919
- [Background] Leslie LK, Wolraich ML. ADHD service use patterns in youth. J Pediatr Psychol. 2007 Jul;32(6):695-710. doi: 10.1093/jpepsy/jsm023. Epub 2007 Jun 7. PMID 17556401
- [Background] Shaw M, Hodgkins P, Caci H, Young S, Kahle J, Woods AG, Arnold LE. A systematic review and analysis of long-term outcomes in attention deficit hyperactivity disorder: effects of treatment and non-treatment. BMC Med. 2012 Sep 4;10:99. doi: 10.1186/1741-7015-10-99. PMID 22947230
- [Background] Pelham WE, Foster EM, Robb JA. The economic impact of attention-deficit/hyperactivity disorder in children and adolescents. J Pediatr Psychol. 2007 Jul;32(6):711-27. doi: 10.1093/jpepsy/jsm022. Epub 2007 Jun 7. PMID 17556402
- [Background] Schoenfeld DA. Sample-size formula for the proportional-hazards regression model. Biometrics. 1983 Jun;39(2):499-503. PMID 6354290
- [Background] Xie H, McHugo G, Drake R, Sengupta A. Using discrete-time survival analysis to examine patterns of remission from substance use disorder among persons with severe mental illness. Ment Health Serv Res. 2003 Mar;5(1):55-64. doi: 10.1023/a:1021759509176. PMID 12602646

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Usual Care Plus Assessment
Started | 112 | 95
1 Month Follow up | 67 | 50
3 Month Follow up | 50 | 43
6 Month Follow up | 33 | 25
Completed | 33 | 25
Not Completed | 79 | 70
Not completed — Lost to Follow-up | 47 | 47
Not completed — Never started ADHD medication | 32 | 23

BASELINE CHARACTERISTICS:
Population: The population under study consists of children under age 18 who presented at 4 clinics in Northern California Kaiser Permanente for ADHD assessment. The study baseline population consists of 207 potentially eligible participants who enrolled and signed consent for the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Usual Care Plus Assessment | Total
Number analyzed (Participants) | 112 | 95 | 207
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 112 | 95 | 207
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.5 (1.9) | 8.5 (1.9) | 8.5 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 27 | 57
  Male | 82 | 68 | 150
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 112 | 95 | 207

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 25% Reduction in SNAP Scores
Description: Outcome measure reported is the number of participants with at least one 25% reduction in SNAP between visits. In treatment of ADHD, the therapeutic dose is defined as a 25% reduction in SNAP IV score between consecutive clinic visits. SNAP is itemized rating scale (Swanson, Nolan, and Pelham-IV Questionnaire) designed to measure ADHD symptoms and severity on a 4 point scale. It is based on DSM IV criteria, and is designed to measure attention deficit hyperactivity disorder (ADHD) and oppositional defiant disorder (ODD) symptoms in children and young adults ages 6-18.
Time Frame: One month, 3 month and six month follow ups
Population: Fifty eight (58) participants completed the study (i.e., had their 6 month follow up appointment) when the study was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Usual Care Plus Assessment
Number analyzed (Participants) | 33 | 25
Participants | 29 | 23

2. Secondary Outcome: ADHD Symptomatology
Description: Outcomes reported are average SNAP IV scores at baseline and 6 monhts. ADHD symptomatology is measured by the Swanson, Nolan and Pelham Teacher and Parent Rating Scale (SNAP-IV), developed by James Swanson, Edith Nolan and William Pelham. We used the 18-item self-report inventory designed to measure attention deficit hyperactivity disorder (ADHD) symptoms in children and young adults. Each question measures the frequency of a variety of symptoms or behaviors.The subscales measure Inattention (9 items) and Hyperactivity/impulsivity (9 items), using 0-3 rating, 0="not at all", 1="just a little", 2="quite a bit", or 3="very much. Each 9-item subscale results in a score in range 0-27. The two subscale scores were averaged to create a single score for the 18-item SNAP.
Time Frame: 6 months post baseline
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Usual Care | Usual Care Plus Assessment
Number analyzed (Participants) | 33 | 25
Score on a scale
  Average SNAP score at baseline | 17.4 (4.8) | 15.0 (4.4)
  Average SNAP score at 6 months | 9.0 (5.6) | 8.6 (5.9)

3. Secondary Outcome: Academic Performance
Description: Academic performance will be measured by student report cards, and converted to a standardized scale
Time Frame: Baseline and Six Months
Population: Academic performance was not measured, as there were a very low number of report cards collected (11 of 25 in Quotient arm and 16 of 33 in UC arm).
Arm/Group | Usual Care | Usual Care Plus Assessment
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

4. Secondary Outcome: Persistence in Care
Description: Update: Outcome measure reported is the # of participants who attended all study follow-up visits.
  Use of pediatric health care services
Time Frame: Baseline to Six Months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Usual Care Plus Assessment
Number analyzed (Participants) | 33 | 25
Participants | 30 | 25

5. Secondary Outcome: Medication Adherence
Description: Update: Outcome reported is number of participants taking medication as prescribed at all study follow up visits.
  Sustained use of ADHD medication
Time Frame: Baseline to six months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Usual Care Plus Assessment
Number analyzed (Participants) | 33 | 25
Participants | 18 | 17

6. Secondary Outcome: Satisfaction With Care
Description: Update: Outcome measure reported is number of participants who responded "very satisfied" with their ADHD care on 5-point Likert scale.
  Likert scale single item measure of how satisfied the pediatric patient's parent was with care received
Time Frame: Six months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Usual Care Plus Assessment
Number analyzed (Participants) | 33 | 25
Participants | 28 | 20

7. Secondary Outcome: Other Health Services Use
Description: Update: Outcome measure reported is number of psychiatric and ED visits during the 6 month follow up period.
  Use of healthcare services outside of pediatrics, including the emergency room and psychiatric services.
Time Frame: Baseline to six months
Measure: Number; unit: visits
Arm/Group | Usual Care | Usual Care Plus Assessment
Number analyzed (Participants) | 33 | 25
visits
  Number of psych visits | 26 | 22
  Number of ED visits | 4 | 2

ADVERSE EVENTS:
Time Frame: 6 months (from baseline to 6 month follow up)
Description: Adverse events were assessed via periodic chart reviews of study participants..
Arm/Group | Usual Care | Usual Care Plus Assessment
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/95
Serious Adverse Events (participants affected / at risk) | 1/112 | 0/95
Other Adverse Events (participants affected / at risk) | 0/112 | 0/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=112) | Usual Care Plus Assessment (N=95)
Ashthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Through chart review, it was discovered one patient was hospitalized due to severe asthma attack. Child has history of asthma, and this episode was likely triggered by URI. Was deemed by DSMB to not be related to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No